CLINICAL TRIAL: NCT04309474
Title: A Randomized, Double-Blind, Placebo-Controlled Proof-of-Concept Study to Assess the Safety and Efficacy of Elezanumab in Acute Ischemic Stroke
Brief Title: A Safety and Efficacy Study of Intravenous (IV) Elezanumab Assessing Change in Neurologic Function in Adult Participants With Acute Ischemic Stroke
Acronym: EAISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M19-148; 2019-003753-29 (EudraCT Number)
Record Dates: First submitted 2020-03-13; First posted 2020-03-16 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; ABT-555; Elezanumab; EAISE
MeSH Terms: conditions — Ischemic Stroke | interventions — elezanumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elezanumab (Experimental): Participants will receive elezanumab 1800 mg
  Interventions: Drug: Elezanumab
- Placebo (Placebo Comparator): Participants will receive placebo for elezanumab
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elezanumab — Intravenous (IV) infusion
  Other Names: ABT-555
  Arms: Elezanumab
Drug: Placebo — Intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
Stroke is one of the leading causes death and major functional disability worldwide. Treatment options for acute stroke are limited with many patients having residual neurologic impairment. The purpose of this study is to evaluate the safety and efficacy of elezanumab and assess change in neurologic function in participants following an acute ischemic stroke.

Elezanumab is an investigational drug being developed for the treatment of acute ischemic stroke. This 52-week study is "double-blinded', which means that neither the participants nor the study doctors will know who will be given elezanumab and who will be given placebo (does not contain treatment drug). Participants will be assigned to one of two groups, called treatment arms. Participants in one arm will receive elezanumab and participants in the other arm will receive placebo. There is a 1 in 2 chance that participants will be assigned to placebo. Approximately 120 subjects will be enrolled in 45 sites worldwide.

Participants will be randomized to elezanumab or placebo by intravenous (IV) infusion within 24 hours of "last known normal" (time when the participant was last known to be without signs and symptoms of the current stroke) and every 4 weeks thereafter for 48 weeks for a total of 13 doses.

There may be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of elezanumab will be checked by medical assessments, blood tests, evaluation of side effects, and completion of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke, supported by acute brain computed tomography (CT) or magnetic resonance imaging (MRI) consistent with the clinical diagnosis.
* Able to randomize within 24 hours of last known normal.
* National Institute of Health Stroke Scale (NIHSS) total score of 7 to 21, inclusive.
* Participants or their legally authorized representative confirms that prior to index stroke, no significant impairment in participant's ability to perform activities of daily living without assistance.

Exclusion Criteria:

* Evidence of severe stroke on imaging based on available acute imaging studies performed under the standard of care.
* Evidence of acute seizure at the onset of index stroke without conclusive imaging of ischemic stroke.
* Evidence of acute myocardial infarction.
* Symptoms are considered likely to resolve within the subsequent few hours (e.g., transient ischemic attack [TIA]).
* Known history prior to randomization of clinically significant medical conditions (other than current acute ischemic stroke) or any other reason, including any physical, psychological, or psychiatric condition that in the investigator's opinion would compromise the safety or interfere with the participant's participation in this study.
* Known medical history of repeated episodes of complex migraine. Participants with history of complex migraine, but with imaging conclusively demonstrating an acute ischemic stroke are still allowed.
* Female who is pregnant, breastfeeding, or considering becoming pregnant during the study or for within 39 weeks (5 half-lives) after the last dose of study drug.
* Known receipt of any investigational product within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug. No current enrollment in another interventional clinical study, including pharmacologic and behavioral interventional studies.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (42):
- United States (22):
  - Mayo Clinic Arizona /ID# 214957, Phoenix, Arizona
  - Long Beach Medical Center /ID# 217210, Long Beach, California
  - Georgetown University Hospital /ID# 216481, Washington D.C., District of Columbia
  - Duplicate_Mayo Clinic /ID# 217567, Jacksonville, Florida
  - Northwestern University Feinberg School of Medicine /ID# 215047, Chicago, Illinois
  - Duplicate_University of Kentucky Chandler Medical Center /ID# 216394, Lexington, Kentucky
  - University of Louisville Hospital /ID# 217569, Louisville, Kentucky
  - Tufts Medical Center /ID# 215053, Boston, Massachusetts
  - University of Mississippi Medical Center /ID# 217587, Jackson, Mississippi
  - St. Luke's Marion Bloch Neuroscience Institute /ID# 215028, Kansas City, Missouri
  - Washington University-School of Medicine /ID# 214526, St Louis, Missouri
  - Hackensack Univ Med Ctr /ID# 218200, Hackensack, New Jersey
  - University of New Mexico School of Medicine /ID# 216827, Albuquerque, New Mexico
  - Columbia University Medical Center /ID# 215122, New York, New York
  - UH Cleveland Medical Center /ID# 215372, Cleveland, Ohio
  - Cleveland Clinic Main Campus /ID# 214635, Cleveland, Ohio
  - The Ohio State University /ID# 215036, Columbus, Ohio
  - Lehigh Valley Health Network /ID# 242446, Allentown, Pennsylvania
  - Thomas Jefferson University Hospital /ID# 215469, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at Houston /ID# 215018, Houston, Texas
  - Baylor Scott & White Medical Center- Temple /ID# 225513, Temple, Texas
  - University of Virginia /ID# 215757, Charlottesville, Virginia
- Australia (2):
  - Duplicate_Royal North Shore Hospital /ID# 239083, St Leonards, New South Wales
  - The Royal Melbourne Hospital /ID# 240178, Parkville, Victoria
- Canada (2):
  - University of Alberta Hospital /ID# 218370, Edmonton, Alberta
  - Hamilton General Hospital /ID# 218970, Hamilton, Ontario
- Japan (5):
  - Fukuoka University Chikushi Hospital /ID# 240629, Chikushino-shi, Fukuoka
  - Fukuoka Wajiro Hospital /ID# 239810, Fukuoka, Fukuoka
  - National Hospital Organization Kagoshima Medical Center /ID# 240021, Kagoshima, Kagoshima-ken
  - Nagano Municipal Hospital /ID# 240622, Nagano, Nagano
  - Yamaguchi Grand Medical Center /ID# 239892, Hohu-shi, Yamaguchi
- South Korea (4):
  - Duplicate_Pusan National University Hospital /ID# 233769, Busan, Busan Gwang Yeogsi
  - Duplicate_CHA University Bundang Medical Center /ID# 233503, Seongnam-si, Gyeonggido
  - Seoul National University Hospital /ID# 233473, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 234241, Seoul, Seoul Teugbyeolsi
- Spain (7):
  - Complejo Hospitalario Universitario A Coruña /ID# 230080, A Coruña, A Coruna
  - Hospital Donostia /ID# 218034, Donostia / San Sebastian, Guipuzcoa
  - OSI Ezkerraldea-Enkarterri-Cruces /ID# 217529, Barakaldo, Vizcaya
  - Hospital Universitario Vall de Hebron /ID# 217087, Barcelona
  - Hospital Universitario La Paz /ID# 216380, Madrid
  - Hospital Universitario Virgen Macarena /ID# 216382, Seville
  - Hospital Universitario Virgen del Rocio /ID# 216339, Seville

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants will receive placebo for elezanumab via Intravenous (IV) infusion.
- Elezanumab: Participants will receive elezanumab 1800 mg via Intravenous (IV) infusion.
Period: Overall Study
Arm/Group | Placebo | Elezanumab
Started (Randomized subjects) | 60 | 61
Treated | 60 | 59
Completed (Completed study treatment) | 39 | 41
Not Completed | 21 | 20
Not completed — Randomized but not treated | 0 | 2
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — Not disclosed | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elezanumab | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Customized [Count of Participants; unit: Participants]
  < 70 years | 27 | 25 | 52
  70 to < 80 years | 18 | 19 | 37
  ≥ 80 years | 15 | 15 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 24 | 56
  Male | 28 | 35 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 53 | 54 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 46 | 45 | 91
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Analysis of the National Institutes of Health Stroke Scale (NIHSS) Total Score Area Under the Curve During the Treatment Period
Description: The National Institutes of Health Stroke Scale (NIHSS) is a neurological examination used to quantitatively measure the severity of acute stroke by evaluating impact of cerebral infarction on level of consciousness, gaze, visual field, facial palsy, motor ability of arm and leg, limb ataxia, sensation, language, dysarthria, and extinction/inattention. Domains are scored on a scale of 0 to 2, 0 to 3, or 0 to 4, for a total range of 0 to 42 points with higher scores indicating impairment.
  The monthly-adjusted AUC of the NIHSS total score for each treatment group was derived using the trapezoidal method and contrasts from a Mixed Model with Repeated Measures (MMRM). Please refer to the formula for AUCi in the Statistical Analysis Plan (SAP) where i = treatment group (placebo, elezanumab) and j = visit during the Treatment Period {Day 1, Day 2-4, Week 4, Week 8, Week 12, Week 24, Week 36, Week 52}.
Time Frame: Day 1 through Week 52
Population: Full Analysis Set
  Note: The AUC for each treatment group, as well as the difference in AUCs (placebo minus elezanumab) and their respective standard errors and confidence intervals are presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Elezanumab
Number analyzed (Participants) | 60 | 59
units on a scale | 3.83 [2.642 to 5.024] | 3.13 [1.938 to 4.317]
Statistical Analysis 1: Comparison: Placebo vs Elezanumab; Test type: Other — A statistical test was not performed; Area under the curve (AUC) = 0.71, 95% CI 2-sided [-0.764 to 2.175] — AUC analyses based on trapezoidal rule using contrast derived from MMRM with stratification factors, treatment, visit, and a treatment by visit interaction included in the model. Posterior probability that the difference in AUC exceeds 0.6 = 0.557

2. Secondary Outcome: Responder Status Based on Modified Rankin Scale (mRS)
Description: The mRS is used to assess participant's disability and functional dependence. It is a 6-point scale ranging from 0 (no symptoms) to 5 (severe disability), with additional rating of 6 if the participant is deceased.
Time Frame: Week 52
Population: Full Analysis Set
  N indicates the number of subjects with non-missing values at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Elezanumab
Number analyzed (Participants) | 46 | 38
Participants | 28 | 29
Statistical Analysis 1: Comparison: Placebo vs Elezanumab; Test type: Other — A statistical test was not performed; Odds Ratio of LS Means = 1.74, 95% CI 2-sided [0.71 to 4.24] — Point estimate for responder rate (defined as having an mRS score of 0, 1, or 2), odds ratio and 95% confidence intervals based on a generalized linear mixed model (GLMM)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 608.5 and 607 days for Placebo and Elezanumab 1800 mg, respectively.
Arm/Group | Placebo | Elezanumab
All-Cause Mortality (participants affected / at risk) | 7/60 | 1/61
Serious Adverse Events (participants affected / at risk) | 23/60 | 18/61
Other Adverse Events (participants affected / at risk) | 52/60 | 49/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Elezanumab (N=61)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC VENTRICULAR THROMBOSIS (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 1 (2) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
MUCOSAL DRYNESS (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
HAEMOPHILUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
PNEUMONIA ASPIRATION (Infections and infestations) | 2 (2) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TROPONIN INCREASED (Investigations) | 0 (0) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYELOPROLIFERATIVE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 1 (1)
BASILAR ARTERY THROMBOSIS (Nervous system disorders) | 1 (1) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 3 (3) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 2 (2) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 2 (3)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
FACIAL PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 1 (1)
HAEMORRHAGIC TRANSFORMATION STROKE (Nervous system disorders) | 2 (2) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 3 (3) | 0 (0)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
PARTIAL SEIZURES (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 1 (1) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (2)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Elezanumab (N=61)
ATRIAL FIBRILLATION (Cardiac disorders) | 8 (10) | 6 (6)
BRADYCARDIA (Cardiac disorders) | 4 (5) | 1 (1)
DRY EYE (Eye disorders) | 3 (3) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 13 (14) | 11 (13)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 4 (4)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 7 (7)
FATIGUE (General disorders) | 3 (3) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 6 (6) | 1 (1)
PERIPHERAL SWELLING (General disorders) | 4 (4) | 0 (0)
PYREXIA (General disorders) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 10 (10) | 5 (5)
URINARY TRACT INFECTION (Infections and infestations) | 11 (16) | 13 (16)
FALL (Injury, poisoning and procedural complications) | 11 (15) | 5 (7)
SKIN LACERATION (Injury, poisoning and procedural complications) | 3 (3) | 4 (6)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (9) | 6 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
DIZZINESS (Nervous system disorders) | 3 (4) | 6 (6)
HAEMORRHAGIC TRANSFORMATION STROKE (Nervous system disorders) | 5 (5) | 7 (7)
HEADACHE (Nervous system disorders) | 10 (11) | 7 (8)
SYNCOPE (Nervous system disorders) | 5 (6) | 1 (1)
ANXIETY (Psychiatric disorders) | 5 (6) | 6 (6)
DEPRESSED MOOD (Psychiatric disorders) | 3 (4) | 4 (6)
DEPRESSION (Psychiatric disorders) | 3 (3) | 5 (5)
INSOMNIA (Psychiatric disorders) | 6 (6) | 10 (10)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 5 (6)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4)
HYPERTENSION (Vascular disorders) | 10 (13) | 4 (4)
HYPOTENSION (Vascular disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT04309474/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT04309474/SAP_001.pdf